CLINICAL TRIAL: NCT00011635
Title: The Effect of Milk Thistle on the Pharmacokinetics of Indinavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010054; 01-CC-0054
Record Dates: First submitted 2001-02-24; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-12

CONDITIONS: HIV Infection; Healthy
Keywords: Caffeine; Cytochrome P 450; Dextromethorphan; Drug Interaction; Metabolism; Drug Metabolism; Healthy Volunteer; Milk Thistle
MeSH Terms: conditions — HIV Infections | interventions — Silymarin; milk-thistle extract

INTERVENTIONS:
Drug: Silymarin (milk thistle)

SUMMARY:
Complementary and alternative medicines are widely used in the HIV-infected population. Recent data have shown serious drug interactions between certain complementary medicines and protease inhibitors. Silymarin (Milk thistle) is a commonly used dietary supplement in HIV-infected patients for treatment of hepatitis or as a hepato-protectant. Data are available suggesting that it may alter cytochrome P4503A4-mediated drug metabolism. To evaluate the effect of milk thistle on the protease inhibitor, indinavir (IDV), ten healthy subjects will receive IDV (Crixivan) alone and in combination with an over-the-counter silymarin preparation. IDV will initially be administered alone at a dose of 800 mg Q8H for four doses and serial samples will be collected for determination of IDV pharmacokinetics after the morning dose on day 2. Subjects will then initiate therapy will milk thistle using a standardized formulation and dose for three weeks after which subjects will then again take 4 doses of IDV and have serial samples collected for IDV plasma concentrations. There will then be a 11-day washout period with no drugs, after which IDV will again be given for 4 doses and samples will be collected evaluate the offset of the effects of milk thistle. To examine the effect of milk thistle on other CYP450 pathways, subjects will receive a single dose of caffeine and dextromethorphan and have urine collected before and after milk thistle, and after the washout period. Indinavir, caffeine, and dextromethorphan concentrations in plasma or urine will be determined using validated HPLC methods. Steady-state noncompartmental parameters of indinavir in the presence and absence of milk thistle will be determined. Pharmacokinetic parameters will be compared using ANOVA that will include factors for a period effect and a treatment effect. Statistical analyses will include calculation of the mean ratio of the AUC in the treatment phases compared to IDV alone and determination of 95% confidence intervals. This study will help define the drug interaction potential of complementary and alternative therapies in HIV-infected patients.

DETAILED DESCRIPTION:
Complementary and alternative medicines are widely used in the HIV-infected population. Recent data have shown serious drug interactions between certain complementary medicines and protease inhibitors. Silymarin (Milk thistle) is a commonly used dietary supplement in HIV-infected patients for treatment of hepatitis or as a hepato-protectant. Data are available suggesting that it may alter cytochrome P4503A4-mediated drug metabolism. To evaluate the effect of milk thistle on the protease inhibitor, indinavir (IDV), ten healthy subjects will receive IDV (Crixivan) alone and in combination with an over-the-counter silymarin preparation. IDV will initially be administered alone at a dose of 800 mg Q8H for four doses and serial samples will be collected for determination of IDV pharmacokinetics after the morning dose on day 2. Subjects will then initiate therapy will milk thistle using a standardized formulation and dose for three weeks after which subjects will then again take 4 doses of IDV and have serial samples collected for IDV plasma concentrations. There will then be an 11-day washout period with no drugs, after which IDV will again be given for 4 doses and samples will be collected evaluate the offset of the effects of milk thistle. To examine the effect of milk thistle on other CYP450 pathways, subjects will receive a single dose of caffeine and dextromethorphan and have urine collected before and after milk thistle, and after the washout period. Indinavir, caffeine, and dextromethorphan concentrations in plasma or urine will be determined using validated HPLC methods. Steady-state noncompartmental parameters of indinavir in the presence and absence of milk thistle will be determined. Pharmacokinetic parameters will be compared using ANOVA that will include factors for a period effect and a treatment effect. Statistical analyses will include calculation of the mean ratio of the AUC in the treatment phases compared to IDV alone and determination of 95% confidence intervals. This study will help define the drug interaction potential of complementary and alternative therapies in HIV-infected patients.

ELIGIBILITY:
Age 18 to 65 years.

Healthy by medical history and physical exam.

No concurrent chronic medications, including oral contraceptives.

Non-smoker or not having smoked for the past 6 months or longer.

Laboratory values within established NIAID guidelines for participation in clinical studies: AST/SGOT less than or equal to 2 times ULN; Serum creatinine less then or equal to ULN; Hemoglobin greater than or equal to 10 g/dl.

Ability to abstain from caffeine containing foods/beverages, ethanol, grapefruit or grapefruit juice and charbroiled foods for 72 hours prior to, and the day of, phenotyping procedures.

Ability to abstain from dextromethorphan-containing over the counter preparations for 72 hours prior to, and the day of, phenotyping procedures.

No concomitant therapy with other inhibitors or inducers of cytochrome P-450 mediated drug metabolism within 30 days of study (including grapefruit juice).

No ingestion of dietary supplements within the past 30 days.

Ability to obtain venous access for sample collection.

No presence of life-threatening or unstable renal, hepatic, cardiovascular, hematologic, neurologic, psychiatric, or respiratory disease or any other condition that may interfere with the interpretation of the study results or not be in the best interests of the patient in the opinion of the investigator.

Patients must not have a positive pregnancy test.

No presence of persistent diarrhea or malabsorption that would interfere with the patient's ability to adequately absorb drugs.

No drug or alcohol use that may impair safety or adherence.

No history of intolerance to milk thistle, indinavir, caffeine, or dextromethorphan preparations.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2001-02; Study Completion 2001-06

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Patterns of use, and perceived efficacy of complementary and alternative therapies in HIV-infected patients
- [Background] Ernst E. Second thoughts about safety of St John's wort. Lancet. 1999 Dec 11;354(9195):2014-6. doi: 10.1016/S0140-6736(99)00418-3. No abstract available. PMID 10636361
- [Background] Eisenberg DM, Davis RB, Ettner SL, Appel S, Wilkey S, Van Rompay M, Kessler RC. Trends in alternative medicine use in the United States, 1990-1997: results of a follow-up national survey. JAMA. 1998 Nov 11;280(18):1569-75. doi: 10.1001/jama.280.18.1569. PMID 9820257